CLINICAL TRIAL: NCT04754685
Title: Assessments of Therapeutic Effects of Platelet-rich Plasma in Knee Osteoarthritis: Possible Role of Inflammatory Cytokines
Brief Title: Platelet-rich Plasma and Synovial Cytokines in Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Mohammed H. Hassan, Associate Professor of Medical Biochemistry, Faculty of Medicine , South Valley University, South Valley University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SVU-QFM-102
Record Dates: First submitted 2021-02-05; First posted 2021-02-15 (Actual); Last update posted 2021-02-15 (Actual); Status verified 2021-02

CONDITIONS: Knee Osteoarthritis
Keywords: Platelet rich plasma; Knee osteoarthritis; MRI Osteoarthritis Knee Score; pain score; synovial fluid; tumor necrosis factor-α; macrophage migration inhibitory factor
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: A prospective study was performed on 90 patients were included and categorized into mild (30 cases, moderate (30 cases) and severe (30 cases) knee OA. Three intra-articular (I.A) injections of PRP, 2 weeks a part, were received. Pain score and MRI Osteoarthritis Knee Score (MOAKS) were assessed. Serial synovial fluid cytokines assays in the form of Tumor necrosis factor-α (TNF-α) and Macrophage migration inhibitory factor (MIF), were performed using commercially available ELISA assay kits. The assays were performed pre-injection (S1), two weeks from the 1st I.A injection and two weeks from the 2nd I.A injection (S3) for all included patients.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mild knee osteoarthritis (Active Comparator): 30 patients had mild knee osteoarthritis
  Interventions: Drug: Intra-articular injection of platelet-rich plasma
- Moderate knee osteoarthritis (Active Comparator): 30 patients had moderate knee osteoarthritis
  Interventions: Drug: Intra-articular injection of platelet-rich plasma
- Severe knee osteoarthritis (Active Comparator): 30 patients had severe knee osteoarthritis
  Interventions: Drug: Intra-articular injection of platelet-rich plasma

INTERVENTIONS:
Drug: Intra-articular injection of platelet-rich plasma — The patient was put in 20 degree flexion in supine position with the knee. Under aseptic conditions, a 21-gage needle was used to inject 5 mL of PRP into the suprapatellar knee joint pouch, using a superolateral method. Local anesthetics were not used. Patients were instructed after the injection to refrain from physical exercise for at least 24 hours but no restriction was specified regarding activities of daily living. Three IA-PRP injections were administered at 2-week intervals. The same physician who was engaged in selecting and testing participants did the injections
  Other Names: PRP injection

SUMMARY:
A prospective study was performed on 90 patients were included and categorized into mild (30 cases, moderate (30 cases) and severe (30 cases) knee OA. Three intra-articular (I.A) injections of PRP, 2 weeks a part, were received. Pain score and MRI Osteoarthritis Knee Score (MOAKS) were assessed. Serial synovial fluid cytokines assays in the form of Tumor necrosis factor-α (TNF-α) and Macrophage migration inhibitory factor (MIF), were performed using commercially available ELISA assay kits. The assays were performed pre-injection (S1), two weeks from the 1st I.A injection and two weeks from the 2nd I.A injection (S3) for all included patients.

DETAILED DESCRIPTION:
Background: Osteoarthritis (OA) is a multifactorial disease that commonly affects the knee. Tumor necrosis factor-α (TNF-α) is able to regulate inflammation in OA. Macrophage migration inhibitory factor (MIF) may be involved in the pathophysiology of arthritis. Platelet-rich plasma (PRP) may reduce pain associated with OA. The current study aimed to assess the possible therapeutic effects of PRP in patients with knee OA of various severities.

Methods: A prospective study was performed on 90 patients were included and categorized into mild (30 cases, moderate (30 cases) and severe (30 cases) knee OA. Three intra-articular (I.A) injections of PRP, 2 weeks a part, were received. Pain score and MRI Osteoarthritis Knee Score (MOAKS) were assessed. Serial synovial fluid cytokines assays in the form of Tumor necrosis factor-α (TNF-α) and Macrophage migration inhibitory factor (MIF), were performed using commercially available ELISA assay kits. The assays were performed pre-injection (S1), two weeks from the 1st I.A injection and two weeks from the 2nd I.A injection (S3) for all included patients.

PRP preparation: The PRP needed for IA injection has been prepared under complete aseptic conditions. In order to avoid the effect of food intake on purified PRP, on the day of injection the patients were instructed to fast for 4 hours before blood collection. Approximately 20 mL of venous blood were drawn from the antecubital vein using an aseptic technique in an effort to avoid irritation and trauma to the platelets. Anti-coagulated blood was obtained in ten extraction tubes (2 mL each), containing sodium citrate. The tubes were then centrifuged at 2100 rpm at room temperature for 8 minutes to separate the blood in each tube into the citrated plasma, the buffy coat and the residual red blood cells ( RBCs) . Using a pipette, the PRP situated just above the selectively precipitated RBCs but not including the buffy coat was carefully aspirated from each tube. In each affected joint, 10-mL PRP samples (from the collected venous blood) were used for IA injection . For each intra-articular injection new fresh PRP samples were made from the patients.

ELIGIBILITY:
Inclusion Criteria:

• All patients have unilateral knee OA

Exclusion Criteria:

* Polyarticular disease.
* Knee arthroscopy in the previous year.
* HA or steroid IA penetration in the preceding 3 months.
* History of infectious disease and autoimmune disorders such as diabetes, rheumatoid arthritis.
* Hematologic diseases (coagulopathy).
* Serious cardiovascular diseases , infections or immunodepression.
* Anticoagulant therapy or an anti-aggregating agent.
* Uuse of non-steroidal anti-inflammatory drugs 2 weeks prior to blood sampling.
* < 10 g / dL of hemoglobin

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-03-14 (Actual)

PRIMARY OUTCOMES:
Changes in Pain Scores in patients with various severities of knee OA following intra-articular injection of PRP at 0, and 2 weeks from the second injection (0,4 weeks). | one year
  Using Visual Analog Scale (VAS) score to assess the pain score in patients with knee osteoarthritis will be done twice , pre-intra-articular injection of PRP and 2 weeks from the second I.A injection of PRP.
  The VAS is a common tool that uses a 10 cm scale for pain intensity measurement, where 0= no pain and 10= unable to move.
Changes in the synovial fluid concentration of the TNF-α and MIF levels folllowing PRP injection, using ELISA assay kits. | one year
  Using ELISA assay kits, synovial fluid concentration of both TNF-α and MIF levels will be measured three times for the same patient (before injection, 2 weeks from the first injection and 2 weeks from the second injection) to explore the serial changes in their levels following IA i injection PRP.
Changes in MRI Osteoarthritis Knee Score (MOAKS) in patients with various severities of knee OA following intra-articular injection of PRP at 0, and 2 weeks from the second injection (0,4 weeks). | one year
  Regarding MRI knee score will be done twice , pre-intra-articular injection of PRP and 2 weeks from the second I.A injection of PRP.
  For assessment of both bone marrow abnormality or patella-femoral cartilage volume (grade I (mild if the lesion involves ˂33% of subregional volume); grade II (Moderate: if the lesion involves 33%- 66% of subregional volume), and grade III (severe: if the lesion involves ˃ 66% of subregional volume).Regarding synovitis: grade 1 (mild or small - fluid continuous in the retropatellar space); grade 2 (Moderate or medium - slight convexity of the suprapatellar bursa), and grade 3 (severe or large - evidence of capsular distension ). Meniscal desintegrity score of 0-3 applied for amount of extrusion in 4 locations: medial meniscus (medial and anterior extrusion) and lateral meniscus (medial and anterior extrusion).
Assess the correlations of synovial fluid TNF-α and MIF levels with both pain and radiological scores will performed among these patients. | one year
  Correlate visual Analog pain Scale and MRI Osteoarthritis Knee Score with the pre-injection cytokine synovial levels and synovial level values 2 weeks from the second IA injection of PRP

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed H Hassan, MD, Principal Investigator — Faculty of Medicine- South Valley University
Locations (1):
- Faculty of Medicine, South valley University, Qina, Qena Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Taniguchi Y, Yoshioka T, Kanamori A, Aoto K, Sugaya H, Yamazaki M. Intra-articular platelet-rich plasma (PRP) injections for treating knee pain associated with osteoarthritis of the knee in the Japanese population: a phase I and IIa clinical trial. Nagoya J Med Sci. 2018 Feb;80(1):39-51. doi: 10.18999/nagjms.80.1.39. PMID 29581613
- [Result] Hunter DJ, Guermazi A, Lo GH, Grainger AJ, Conaghan PG, Boudreau RM, Roemer FW. Evolution of semi-quantitative whole joint assessment of knee OA: MOAKS (MRI Osteoarthritis Knee Score). Osteoarthritis Cartilage. 2011 Aug;19(8):990-1002. doi: 10.1016/j.joca.2011.05.004. Epub 2011 May 23. PMID 21645627
- [Result] Katz J, Melzack R. Measurement of pain. Surg Clin North Am. 1999 Apr;79(2):231-52. doi: 10.1016/s0039-6109(05)70381-9. PMID 10352653